CLINICAL TRIAL: NCT02446262
Title: Neural and Psychological Mechanisms of Pain Perception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 150132; 15-AT-0132
Record Dates: First submitted 2015-05-14; First posted 2015-05-18 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01-05

CONDITIONS: Pain; Normal Physiology; Healthy Volunteers
Keywords: Pain; Visual Analogue Pain Scale; Placebo; Affective Neuroscience; Functional Magnetic Resonance Imaging (fMRI)
MeSH Terms: conditions — Pain | interventions — Neuropsychological Tests

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Substudy 1: Instructed subjects (Other): Participants are instructed about outcomes
  Interventions: Behavioral: Instructions
- Substudy 1: Uninstructed subjects (Other): Participants learn through experience
  Interventions: Behavioral: Instructions
- Substudy 2: heat group (Other): Participants learn about heat outcomes through conditioning
  Interventions: Behavioral: Thermal Pain
- Substudy 2: salt group (Other): Participants learn about salt outcomes through conditioning
  Interventions: Behavioral: Thermal Pain
- Substudy 2: sugar group (Other): Participants learn about sugar outcomes through conditioning
  Interventions: Behavioral: Thermal Pain
- Substudy 3: healthy volunteers (No Intervention): All participants experience all outcomes, within subjects designs
- Substudy 4: healthy volunteers (Other): Participants are instructed to attend toward or away from the stimulus
  Interventions: Behavioral: Attention
- Substudy 5: healthy volunteers (Other): Participants experience both placebo and cue-based expectations within subjects
  Interventions: Behavioral: Placebo instructions

INTERVENTIONS:
Behavioral: Instructions — In sub-study 1, half the participants are instructed about outcomes, half learn through experience.
  Arms: Substudy 1: Instructed subjects; Substudy 1: Uninstructed subjects
Behavioral: Attention — In sub-study 4, participants learn about outcomes and we manipulate attention toward or away from the pain.
  Arms: Substudy 4: healthy volunteers
Behavioral: Thermal Pain — In sub-studies 2 and 3, participants are exposed to thermal stimuli and/or tastants (sugar water, salt water, neutral rinse) and we are measuring how learning varies based on the type of outcome.
  Arms: Substudy 2: heat group; Substudy 2: salt group; Substudy 2: sugar group
Behavioral: Placebo instructions — In sub-study 5, we test whether placebo effects and expectancy cues modulate pain through similar mechanisms.
  Arms: Substudy 5: healthy volunteers

SUMMARY:
Background:

- Painful stimuli cause changes in a network of brain regions called the "Pain Matrix." But most of these regions respond to many other stimuli, not just pain. Researchers want to understand how different factors influence pain. They want to test what happens when people expect different levels of pain and receive treatments that can modify pain. They want to see if these factors influence decisions about pain and how the body responds to it. They also want to compare pain with responses like taste and vision.

Objectives:

- To better understand how pain and emotions are processed and influenced by psychological factors.

Eligibility:

- Healthy volunteers ages 18-50.

Design:

* This study requires 1 to 2 clinic visits that last 1 to 3 hours.
* Participants will be screened with medical history and physical exam.
* Some participants will have one or more magnetic resonance imaging (MRI) scans of their brain. For MRI, participants will lie on a table that slides in and out of a cylinder. The scanner makes loud knocking noises. They will get earplugs.
* Participants heart activity will be recorded with electrocardiogram. Their pulse, sweating, and breathing will be monitored.
* Some participants will take a taste test. Others may perform simple tasks. Others may receive pain in their arm, leg, or hand. The pain will come from heat or electric shocks. Others may judge pain using a topical pain-relieving cream. Some of these tests may be given during MRI.
* Participants will fill out questionnaires.
* The study will last 3 years.

DETAILED DESCRIPTION:
Objective

Pain is one of the most important signals for an organism s survival. The pathways that transfer noxious input from the periphery to the central nervous system are highly conserved across human and animal models. In humans, the ultimate experience of pain is also highly influenced by psychological factors. For example, the placebo effect leads to robust pain relief and can influence responses to noxious stimuli in the human brain. However, the psychological and neurobiological mechanisms by which psychological factors influence pain remain largely unknown.

Pain can be modulated by explicit beliefs about treatments, prior experience and learning, interpersonal processes that support the patient-provider relationship, and contextual factors related to the treatment environment. In the proposed series of experiments, we will systematically investigate the neural and psychological mechanisms that mediate the effects of these factors on acute pain. We will focus on expectations, attention, emotion, conditioning/associative learning, and social factors. These experiments will principally use functional magnetic resonance imaging (fMRI) and psychophysiological measurements, as well as behavioral assays and self-reports. We will examine the effects of different types of pain-related expectations on decisions about pain as well as responses in the brain and periphery. We will also compare acute pain with other hedonic and perceptual processes. This will allow us to distinguish processes that are unique to pain perception from those that are not specific to pain, such as processes involved in perception and decision-making across domains.

Together, the proposed series of experiments aim to elucidate the psychological, neurobiological, and physiological mechanisms that modulate pain. This, in turn, can identify targets for pain treatment and inform mechanistic studies of altered pain processing in clinical populations.

Study Population

We plan to recruit 500 healthy volunteers between age 18 and 50.

Design

The aim of the proposed series of experiments is to understand how expectations, attention, and emotion influence acute pain. We will manipulate expectations about noxious stimuli using associative learning and verbal instructions, in both within-subjects and between-groups designs. We will measure decisions about pain experience (self-report) as well as neural and physiological responses to noxious stimuli that cause pain. We will combine computational modeling with advanced neuroimaging analyses to isolate the neural and psychological mechanisms that mediate the effects of expectations, attention, and emotion on subjective pain. To determine the specificity of these mechanisms, we will compare acute pain modalities (e.g., thermal pain versus shock-induced pain), and we will contrast pain with other hedonic and perceptual domains (e.g., taste).

Outcome measures

Dependent variables for all experiments will include decisions about pain and/or other percepts (e.g., sweetness of a taste) measured with visual analogue scales, reaction time, physiological responses (e.g., skin conductance, pupil dilation), and/or BOLD activation in regions of interest. We are specifically interested in processes within the network of regions known to be involved in pain processing (pain-processing network, PPN), as well as responses in the prefrontal cortex (PFC), ventral striatum (VS), and amygdala. We hypothesize that nociceptive stimuli and pain ratings will be associated with unique patterns of activation within the PPN, whereas responses in regions associated with value, executive function, and decision-making will be common across outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy
* Between 18 and 50 years old
* Fluent in English
* Able to provide written informed consent.

EXCLUSION CRITERIA (all sub-studies):

* Unable to comply with study procedures or follow-up visits.
* Has a major medical condition or medical history that in a clinician's assessment could affect heat sensitivity, pain thresholds, or ability to comply with study procedures. This may include cardiovascular, autonomic, or neurological conditions, including stroke, blindness, deafness, a history of brain damage, or a chronic systemic disease (e.g., diabetes).
* Has a current mood disorder, anxiety disorder, or substance use disorder, or has a history of psychosis, hospitalization for a mental health condition, or recurrent psychiatric episodes.
* Has a medical condition that in a clinician's assessment might affect somatosensation (e.g., Raynaud s disease, peripheral neuropathy, or circulatory disorder).
* Has a current chronic pain condition or has had chronic pain in the past (painful condition lasting more than six months).
* Has a dermatological condition affecting the testing region such as scars, burns, or recent tattoos that might influence cutaneous sensibility.
* Regular use of prescription medication that has a significant effect on pain or heat perception. Excluded medications include central-acting agents such as opiates (morphine, tramadol), antidepressants (amitriptyline, duloxetine, milnacipran), anticonvulsants (gabapentin, pregabalin), anxiolytics (barbituates, benzodiazepines), hypnotics (zolpidem, sodium oxybate), antipsychotics (valproate, lithium, olanzapine), antimigraine agents (sumatriptan, ergotamine), and muscle relaxants (cyclobenzaprine, carisoprodol). Use of analgesic medications, such as non-steroidal anti-inflammatories, salicylates, and acetaminophen, taken on an "as needed" basis is acceptable as long as the last dose taken was within 5 half-lives of testing.
* Is pregnant.
* NIH staff member who is a subordinate/relative/co-worker of any investigator on the protocol.

EXCLUSION CRITERIA (fMRI sub-studies):

* Individuals with conditions that could pose a risk relating to the safety of the fMRI procedure or pain stimulation will be excluded from the MRI portion of the protocol, but may participate in the non-fMRI sessions (with the exception of pregnant women). Such conditions include:

  * Those with ferromagnetic metal in the cranial cavity or eye, e.g. aneurysm clip, implanted neural stimulator, cochlear implant, ocular foreign body.
  * Those with an abnormality on a structural MRI.
  * Those with an implanted cardiac pacemaker or auto-defibrillator.
  * Those with an insulin pump.
  * Those with irremovable body piercing.
  * Pregnant women (based on urine test completed within 24 hours prior to scan).
* Individuals who are left-handed (based on self-report or score on handedness questionnaire) will be excluded from fMRI substudies.

EXCLUSION CRITERIA (placebo analgesia sub-studies):

-Participation in an NIH study of analgesia, as gleaned from CRIS.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-06-11 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Physiological responses (heart rate, skin conductance, respiration, pupil dilation, eye gaze position) | During the study visit in response to painful and non-painful stimuli.
  In behavioral and fMRI experiments, we measure autonomic responses in anticipation and response to painful and non-painful stimuli using non-invasive measures.
Pain perception (pain ratings) | During the study visit in response to painful stimuli.
  Substudies of pain collect pain ratings using a visual analogue scale, either verbally or via computer.
BOLD response in brain regions of interest measured using fMRI | During the study visit in response to painful and non-painful stimuli.
  FMRI substudies proceed following behavioral substudies. We measure brain responses in anticipation and response to painful and non-painful stimuli.

SECONDARY OUTCOMES:
Questionnaire measures (e.g. State-trait anxiety index, Fear of Pain questionnaire, Intolerance of Uncertainty questionnaire, McGill Pain Questionnaire) | Trait measures are collected during initial screening visit ; State measures are collected on every visit
  Personality measures that have been linked with pain and emotion will be tested as moderators of effects on the above outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Y Atlas, Ph.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We will share deidentified data only as per language in the protocol.

REFERENCES:
- [Derived] Atlas LY, Dildine TC, Palacios-Barrios EE, Yu Q, Reynolds RC, Banker LA, Grant SS, Pine DS. Instructions and experiential learning have similar impacts on pain and pain-related brain responses but produce dissociations in value-based reversal learning. Elife. 2022 Nov 1;11:e73353. doi: 10.7554/eLife.73353. PMID 36317867
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-AT-0132.html